CLINICAL TRIAL: NCT06608173
Title: Development and Evaluation of a Multi-media Training Program for Elementary School Bullying and Abuse Prevention: radKIDS 2.0
Brief Title: Evaluation of radKIDS 2.0, a Multi-media Training Program for Elementary School Bullying and Abuse Prevention
Acronym: radKIDS2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saavsus, Inc. (Other)
Collaborators: Oregon Research Institute (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R43MD015695 (NIH); R43MD015695 (NIH)
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Self Esteem; Self Efficacy; Knowledge
Keywords: radKIDS; school-based intervention; bullying; victimization; self-esteem; self-efficacy; safety knowledge; prevention
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Classrooms randomly assigned to this arm will receive instruction as usual, with no intervention
- radKIDS program (Experimental): This is the intervention arm, with the radKIDS2.0 program delivered across 20 weeks.
  Interventions: Behavioral: radKIDS2.0 Safety and Empowerment Education Program

INTERVENTIONS:
Behavioral: radKIDS2.0 Safety and Empowerment Education Program — radKIDS® uses activity-based skill training to help elementary aged children develop personal safety boundaries, critical thinking skills for responding to threats of danger, age-appropriate coping strategies for dealing with current and past victimization, self-assertiveness and physical skills for self-defense, communication skills for reporting incidences to parents/adults, and increasing child self-worth-the program's cornerstone for personal safety and healthy development for elementary students.
  Arms: radKIDS program

SUMMARY:
The goal of this clinical trial is to evaluate an adapted version of the radKIDS® Personal Empowerment and Safety Education Program in randomly assigned 4th grade classrooms.

The primary hypothesis is that students in the radKIDS study arm will have significantly higher growth in safety knowledge, safety skill self-efficacy, confidence in help-seeking and in maintaining personal safety, and self-esteem compared to classrooms in the business as usual condition.

At the student level, researchers will compare 4th grade students in classrooms randomized to receive the radKIDS program to those in classrooms receiving their regular instruction.

Student participants will complete two surveys a few months apart assessing safety knowledge, self-efficacy, and self-esteem. In the radKIDS2.0 arm, students will receive the radKIDS program between the two surveys. In the control arm, students will receive instruction as usual.

DETAILED DESCRIPTION:
Child victimization and injury continue to be major public health challenges, jeopardizing the healthy development of millions of American children every day. Child victimization by peers is linked to poorer mental health in later childhood and adolescence, impacting school outcomes due to higher absenteeism, reduced classroom attentiveness, increased school drop-out, and greater risk for substance abuse, delinquency, and violent behavior. Most successful bullying prevention programs do not align with nationally recommended safety guidelines deemed essential for effectively protecting children from victimization and violence. The radKIDS® Personal Empowerment and Safety Education Program is a school-based program developed in response to these national recommendations. radKIDS® uses activity-based skill training to help elementary aged children develop personal safety boundaries, critical thinking skills for responding to threats of danger, age-appropriate coping strategies for dealing with current and past victimization, self-assertiveness and physical skills for self-defense, communication skills for reporting incidences to parents/adults, and increasing child self-worth-the program's cornerstone for personal safety and healthy development for elementary students. To effectively bring the radKIDS® program to more schools across the country, the National Institute on Minority Health and Health Disparities funded this study to adapt the radKIDS® instructor training and student instruction into a blended online/in-person instructor training and instructional delivery system. To evaluate this new instructor training model, the investigators are inviting 40 schools to participate in a randomized trial, with one 4th grade classroom per school participating in the study. Participating classrooms will be randomly assigned, with half of the classrooms getting the radKIDS® program, and half in the "control" condition, receiving instruction as usual. All participating students will complete two surveys a few months apart, assessing growth in knowledge, safety skill self-efficacy, confidence in help-seeking and in maintaining personal safety, and self-esteem. For schools receiving the program, instructors will be trained with the newly adapted curriculum, and will rate the usability and acceptability of the program. If the modified program is effective and practical for use in schools, wide-spread implementation of radKIDS® could have a large impact on public health by decreasing incidents and risks of victimization and reducing child trauma due to preventable violence, abuse, and injury.

ELIGIBILITY:
Inclusion Criteria:

* A student in a participating 4th grade class
* Able to read and understand English
* Able to understand the study
* Able to assent to participate

Exclusion Criteria:

* Not a student in a participating 4th grade class

Ages: 9 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Piers-Harris Self-Concept Scale | Asked twice, at baseline and about three months after baseline
  Provides a complete picture of self-concept using a simple yes-or-no response format. Students will complete three sub-scales: (1) Happiness and Satisfaction (10 items), (2) Freedom from Anxiety (14 items), and (3) Behavioral Adjustment (14 items). Response options are No = 1 and Yes = 2. Items will be scored and summed such that a higher score indicates a higher self-concept. The summed score range on the Happiness and Satisfaction sub-scale is 10 (min) to 20 (max) and the summed score range on both the Freedom from Anxiety and Behavioral Adjustment sub-scales are 14 (min) to 28 (max).
radKIDS Safety Knowledge | This is done by students twice, at baseline and about three months later.
  The investigators developed this survey to assess student safety knowledge. It consists of 15 safety knowledge questions in a multiple choice format. There is one correct answer to each question, with higher scores indicating more safety knowledge. The correct number of items will be summed, divided by 15, and multiplied by 100 to reflect the percent of items answered correctly. The scores can range from 0 to 100.
Self-efficacy with safety skills | This survey is done twice, once at baseline and once about 3 months later.
  The investigators adapted a self-efficacy scale to apply to child safety skills. Self-efficacy reflects confidence in the ability to exert control over ones own motivation, behavior, and social environment. This scale has 12 items with response options from 1 = Not well at all to 5 = Very well. A mean score will be computed with a possible range of 1 to 5, with higher scores indicating more self-efficacy.
Child Rosenberg Self-esteem Scale | This is done twice, at baseline and about three months later.
  This 10 item self-esteem scale is validated for children ages 7-12 and assesses a positive or negative attitude toward the self. Response options are from 1 - definitely not true, to 4, very true. The investigators will compute a mean score such that higher scores indicate higher self-esteem. The scores can range from 1 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Johnson-Shelton, PhD, Principal Investigator — Saavsus, Inc.
Locations (2):
- United States (2):
  - Saavsus, Inc., Eugene, Oregon
  - Oregon Research Institute, Springfield, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Study data deposited in openICPSR will be available to the research community free of charge and in perpetuity. Study data will be findable by searching for the project title on the openICPSR database.
Supporting Information: Study Protocol, ICF
Time Frame: It will be available within one year of the end of this study, by August 31, 2026. It will be available in perpetuity.
Access Criteria: It will be made publicly available in the openICPSR database, with open access.